CLINICAL TRIAL: NCT02726607
Title: Adapting the HITSystem to Support Prevention of Mother-to-child HIV Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenya Medical Research Institute (Other); Global Health Innovations (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sarah Kessler, PhD, MPH, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002009; R34MH107337-01 (NIH)
Record Dates: First submitted 2016-03-24; First posted 2016-04-01 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: Prevention of mother-to-child transmission (PMTCT); Kenya; HITSystem 2.0; retention through PMTCT cascade of care; Early Infant Diagnosis; eHealth system-level intervention

STUDY DESIGN:
Intervention Model Description: We employed a matched randomized pilot study design in two government hospitals; one randomized to receive the HITSystem 2.0 intervention while the other maintained standard of care PMTCT services.
Oversight: Data Monitoring Committee: No

ARMS (2):
- HITSystem 2.0 (Experimental): Pregnant women who are eligible for PMTCT services will be enrolled in the HIV Infant Tracking System 2.0 (HITSystem 2.0) intervention during their first PMTCT appointment and followed until 12 weeks postpartum.
  Interventions: Behavioral: HIV Infant Tracking System (HITSystem) 2.0
- Standard of PMTCT Care (Active Comparator): Pregnant women who are eligible for PMTCT services will receive standard of care PMTCT services at the control hospital. The records of women enrolled during their first PMTCT appointment will be used to assess outcomes during the same follow-up period.
  Interventions: Behavioral: Standard of PMTCT care

INTERVENTIONS:
Behavioral: HIV Infant Tracking System (HITSystem) 2.0 — The HITsystem 2.0 intervention will be designed to: (1) utilize electronic prompts to notify providers and program managers when actions are required, and (2) send text messages to women's mobile phones to (a) motivate adherence to medication, (b) remind women of antenatal (ANC) appointments and medication refills, (c) prompt preparation for a hospital delivery, and (d) support early infant testing. Given advancements in the approach and protocols for care, HITSystem 2.0 will continue to engage mothers and encourage postnatal medication adherence. The researchers will design HITSystem 2.0 to integrate seamlessly into the existing HITSystem to link PMTCT and early infant diagnosis (EID) services through one coordinated system-level intervention.
  Arms: HITSystem 2.0
Behavioral: Standard of PMTCT care — Pregnant women enrolled in PMTCT services at the control site will receive the current standard of PMTCT care and will not be enrolled in the HITSystem 2.0.
  Other Names: no HITSystem 2.0 intervention
  Arms: Standard of PMTCT Care

SUMMARY:
The purpose of this study is to modify the HITSystem to engage and retain HIV+ pregnant women before, during and after delivery and evaluate the HITSystem impact on prevention of mother-to-child transmission (PMTCT) related behaviors and outcomes. HITSystem 2.0 intervention will support a range of PMTCT outcomes including retention in care, ART adherence, and integration of maternal and pediatric HIV services in low-resource settings.

DETAILED DESCRIPTION:
The study will be conducted in three phases:

Phases 1: The researchers will conduct formative research (focus groups and interviews) with HIV+ pregnant women and PMTCT providers to customize communication strategies for text messaging and inform patient flow and optimal implementation across the various PMTCT-related services at the intervention site.

Phase 2: The researchers will design and refine the HITSystem 2.0 technical components to support PMTCT outcomes guided by clinical content experts, technology analysts, and findings from Phase 1.

Phase 3: The researchers will implement HITSystem 2.0 at one hospital over an 18 month period, and compare targeted PMTCT outcomes to those at a matched control hospital.

The study will be conducted at two government hospitals in Kenya. HIV+ pregnant women will be enrolled in the HITSystem 2.0 at Kapsabet Hospital. HIV+ pregnant women receiving the current standard of PMTCT care at Nandi Hills Hospital will be the comparison group.

ELIGIBILITY:
Phase 3

Inclusion Criteria:

* HIV+ pregnant women
* Present for first PMTCT appointment at one of the study Hospitals
* Own or have reliable access to mobile phone

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Complete PMTCT retention | first PMTCT visit during pregnancy to the return of the infant's first HIV DNA PCR test result by 12 weeks postnatal
  The primary outcome is retention (complete or incomplete), measured from first PMTCT appointment until HIV status determination of the HIV-exposed infant at 12 weeks postnatal. This aggregate outcome includes completion of several intermediate outcomes throughout the PMTCT cascade of care, including: ART initiation (if not already on ART at time of pregnancy) (Yes/No), attendance at PMTCT appointments (Yes/No), a hospital delivery (Yes/No), infant enrollment in EID prior to hospital discharge (Yes/No), infant blood sample collected and HIV DNA PCR test result obtained (Yes/No). Complete retention requires completion of all of these steps.

SECONDARY OUTCOMES:
Duration of PMTCT Retention | Date of first PMTCT appointment through date of last PMTCT service. Final eligible service is date of infant HIV PCR test.
  The mean (sd) duration of PMTCT retention (number of weeks from date of PMTCT enrollment to date of last documented PMTCT service).
Infant HIV status | Results obtained by 12 weeks postnatal
  Result of infant HIV DNA Polymerase Chain Reaction (PCR) test: HIV-positive, HIV-negative, indeterminate, unknown, missing
Number of antenatal PMTCT appointments attended | First antenatal PMTCT appointment through delivery date
  The mean (sd) number of ANC appointments attended, and the proportion of women who received the recommended 4 or more antenatal appointments prior to delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah F Kessler, PhD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (3):
- University of Kansas Medical Center, Kansas City, Kansas, United States
- Kenya (2):
  - Bungoma County Hospital, Bungoma, Nandi
  - Kapsabet Hospital, Kapsabet, Nandi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finocchario-Kessler S, Maloba M, Brown M, Gautney B, Goggin K, Wexler C, Mabachi N, Odeny B, Lagat S, Koech S, Dariotis JK, Odeny TA. Adapting the HIV Infant Tracking System to Support Prevention of Mother-to-Child Transmission of HIV in Kenya: Protocol for an Intervention Development Pilot Study in Two Hospitals. JMIR Res Protoc. 2019 Jun 8;8(6):e13268. doi: 10.2196/13268. PMID 31199305
- [Result] Mabachi NM, Brown M, Sandbulte M, Wexler C, Goggin K, Maloba M, Finocchario-Kessler S. Using a Social Support Framework to Understand How HIV Positive Kenyan Men Engage in PMTCT/EID Care: Qualitative Insights From Male Partners. AIDS Behav. 2020 Jan;24(1):18-28. doi: 10.1007/s10461-019-02451-6. PMID 30877581